CLINICAL TRIAL: NCT05716763
Title: Comparative Randomized, Single Dose, Two-Way Crossover Open Label Study To Determine The Bioequivalence Of 5 mg/mL Tramadol Hydrochloride Oral Solution (08P1902F0) Relative To Contramal® (100 mg/mL Oral Solution) After An Oral Administration
Brief Title: Bioequivalence of IMP 08P1902F0 Relative to Contramal® (100 mg/mL Oral Solution)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unither Pharmaceuticals, France (Industry)
Collaborators: International Pharmaceutical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UP-CLI-2021-001
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tramadol; Solutions

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, single dose, two-sequence, two-period crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol hydrochloride 5mg/mL oral solution (IMP 08P1902F0) (Experimental)
  Interventions: Drug: Tramadol Hydrochloride 5 MG/ML Oral Solution
- Tramadol hydrochloride 100mg/mL oral solution (Contramal(r)) (Active Comparator)
  Interventions: Drug: Tramadol Hydrochloride 100 MG/ML Oral Solution (Contramal(r))

INTERVENTIONS:
Drug: Tramadol Hydrochloride 5 MG/ML Oral Solution — 50mg (10mL) single dose
  Arms: Tramadol hydrochloride 5mg/mL oral solution (IMP 08P1902F0)
Drug: Tramadol Hydrochloride 100 MG/ML Oral Solution (Contramal(r)) — 50mg (20 drops) single dose
  Arms: Tramadol hydrochloride 100mg/mL oral solution (Contramal(r))

SUMMARY:
This study aims to demonstrate the bioequivalence between the formulation of 5 mg/mL Tramadol Hydrochloride Oral Solution (08P1902F0) Relative to the reference product Contramal® (100 mg/mL Oral Solution).

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female human subjects, age 18-50 years
* Body mass index between 18.5-30 Kg/m²
* Subject with normal findings
* Willingness to follow the protocol requirements

Exclusion Criteria:

* History of hypersensitivity to tramadol hydrochloride
* Significant history of asthma, thyrotoxicosis, tumours, peptic or gastric ulcer, gastrointestinal malabsorption or haemorrhage in the gastro-intestinal tract, sinusitis, pharyngitis, renal disorder (impaired renal function), hepatic disorder (impaired hepatic function), cardiovascular disorder (ex. severe heart failure), neurological disease such as epilepsy, haematological disorders or diabetes, psychiatric, dermatologic or immunological disorders
* Presence of any clinically significant results from laboratory tests,
* lactating female or woman of childbearing potential unwilling to use an effective contraception

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Majdi Abu Awida, M.D, Principal Investigator — IPRC
Locations (1):
- IPRC reserach site facility, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: cross-over study.
Groups:
- Tramadol HCl 5mg/mL Oral Solution IMP08P1902F0 Then Tramadol HCl 100mg/mL Oral Solution Contramal(r): Participants first received Tramadol Hydrochloride 5 MG/ML Oral Solution: 50mg (10mL) single dose (IMP 08P1902F0) manufactured by Unither Liquid Manufacturing in a fasting state. After a washout period of 1 week, they received Tramadol HCl 100mg/mL oral solution Contramal(r) manufactured by Grunenthal GmbH in a fasting state
- Tramadol HCl 100mg/mL Oral Solution Contramal(r) Then Tramadol HCl 5mg/mL Oral Solution IMP08P1902F0: Participants first received Tramadol HCl 100mg/mL oral solution Contramal(r) manufactured by Grunenthal GmbH in a fasting state. After a washout period of 1 week, they received Tramadol Hydrochloride 5 MG/ML Oral Solution: 50mg (10mL) single dose (IMP 08P1902F0) manufactured by Unither Liquid Manufacturing in a fasting state.
Period: Period I
Arm/Group | Tramadol HCl 5mg/mL Oral Solution IMP08P1902F0 Then Tramadol HCl 100mg/mL Oral Solution Contramal(r) | Tramadol HCl 100mg/mL Oral Solution Contramal(r) Then Tramadol HCl 5mg/mL Oral Solution IMP08P1902F0
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Period II
Arm/Group | Tramadol HCl 5mg/mL Oral Solution IMP08P1902F0 Then Tramadol HCl 100mg/mL Oral Solution Contramal(r) | Tramadol HCl 100mg/mL Oral Solution Contramal(r) Then Tramadol HCl 5mg/mL Oral Solution IMP08P1902F0
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol HCl 5mg/mL Oral Solution IMP08P1902F0 Then Tramadol HCl 100mg/mL Oral Solution Contramal(r) | Tramadol HCl 100mg/mL Oral Solution Contramal(r) Then Tramadol HCl 5mg/mL Oral Solution IMP08P1902F0 | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6.6) | 29 (7.3) | 27 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Jordan | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Tramadol Hydrochloride for the Test and the Reference Products
Description: The maximum concentration in plasma among observed concentrations at pre-specified time points
Time Frame: predose, 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
Number analyzed (Participants) | 24 | 24
ng/mL | 139.65 (53.01) | 123.90 (36.02)

2. Primary Outcome: AUC0-t of Tramadol Hydrochloride for the Test and the Reference Products
Description: The area under the plasma concentration versus time curve from time 0 to the last measured concentration
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
Number analyzed (Participants) | 24 | 24
ng*h/mL | 902.01 (339.22) | 812.63 (301.24)

3. Secondary Outcome: AUC0-infinity of Tramadol Hydrochloride for the Test and the Reference Products
Description: The area under the plasma concentration versus time curve from time 0 to to infinite time
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
Number analyzed (Participants) | 24 | 24
ng*h/mL | 965.92 (385.19) | 873.74 (344.86)

4. Secondary Outcome: Kel of Tramadol Hydrochloride for the Test and the Reference Products
Description: The elimination rate constant
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
Number analyzed (Participants) | 24 | 24
L/h | 0.1344 (0.04) | 0.1294 (0.03)

5. Secondary Outcome: Tmax of Tramadol Hydrochloride for the Test and the Reference Products
Description: Time of the maximum measured plasma concentration. Determined directly from the plasma concentration-time curve. If the maximum value occurs at more than one time point, tmax is defined as the first time point with this value.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: h
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
Number analyzed (Participants) | 24 | 24
h | 1.5 [0.5 to 2.5] | 1 [0.5 to 2.5]

6. Secondary Outcome: T1/2 of Tramadol Hydrochloride for the Test and the Reference Products
Description: Plasma Elimination Half-Life
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
Number analyzed (Participants) | 24 | 24
h | 5.48 (1.33) | 5.71 (1.48)

7. Secondary Outcome: Number of Treatment-related Adverse Events
Description: Occurence and severity of adverse events (serious and non serious adverse events)
Time Frame: Day 1 to Day 11 (end of study)
Measure: Number; unit: adverse events
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
Number analyzed (Participants) | 24 | 24
adverse events | 0 | 0

8. Other Pre Specified Outcome: Palatability Questionnaire
Description: 5 point scale: from 1 : very bad after taste to 5 : very good after taste
Time Frame: 0 and 2 minutes
Measure: Number; unit: percentage of participant
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
Number analyzed (Participants) | 24 | 24
percentage of participant
  very bad taste at 0 min | 4.17 | 4.17
  bad taste at 0 min | 12.5 | 33.33
  no taste at 0 min | 0 | 0
  good taste at 0 min | 66.67 | 54.17
  very good taste at 0 min | 16.67 | 8.33
  Very bad after taste at 2 min | 0 | 4.17
  bad after taste at 2 min | 4.17 | 29.17
  no after taste at 2 min | 4.17 | 20.83
  good after taste at 2 min | 66.67 | 41.67
  very good after taste at 2 min | 25 | 4.17

ADVERSE EVENTS:
Time Frame: Before dosing and 24 hours after each intervention administration, up to 2 days total
Arm/Group | Tramadol Hydrochloride 5mg/mL Oral Solution (IMP 08P1902F0) | Tramadol Hydrochloride 100mg/mL Oral Solution (Contramal(r))
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study are Unither-Pharmaceuticals proprietary and cannot be published or presented in any scientific meeting without any agreement from the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT05716763/Prot_SAP_000.pdf